CLINICAL TRIAL: NCT05791474
Title: A Phase Ia Trial of ATI-2231 in Advanced Solid Tumor Malignancies
Brief Title: ATI-2231 in Advanced Solid Tumor Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Washington University School of Medicine (Other)
Collaborators: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202306048
Record Dates: First submitted 2023-01-31; First posted 2023-03-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumor; Advanced Solid Tumor Malignancies
Keywords: MK2 inhibitor; ATI-2231

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATI-2231 monotherapy dose escalation (Experimental): * Patients will receive single agent ATI-2231 at assigned dose levels (n=3-6 per dose level). Starting dose of 20 mg by mouth twice per day.
  * Each cycle is 21 days
  Interventions: Drug: ATI-2231

INTERVENTIONS:
Drug: ATI-2231 — Provided by Aclaris Therapeutics, Inc.

SUMMARY:
The purpose of this first-in-human study is to test ATI-2231 in advanced solid tumor malignancies with the goal of establishing the recommended Phase II dose of ATI-2231.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven advanced solid tumor malignancy including head and neck cancer, non-small cell lung cancer, gastrointestinal adenocarcinoma, pancreatic adenocarcinoma, prostate cancer, bladder cancer, and breast cancer.
* Eligible patients must have an advanced solid malignancy above, for which standard curative or palliative therapies do not exist or are no longer effective.
* Measurable or non-measurable but evaluable disease by RECIST v 1.1.
* Patients must have archival tissue sample available from prior metastatic biopsy. If no tissue is available, patient may still be able to enroll with PI approval.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Life expectancy of at least 12 weeks.
* Adequate bone marrow and organ function as defined below:

  * Leukocytes ≥ 3 K/cumm
  * Absolute neutrophil count (ANC) ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Total bilirubin ≤ 1.5 x IULN (unless patient has known Gilberts disease)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 60 mL/min by Cockcroft-Gault
* The effects of ATI-2231on the developing human fetus are unknown. For this reason, women of childbearing potential and men who are heterosexually active must agree to use adequate contraception as specified in the protocol. Contraception should continue for 1 month (for women) or 3 months (for men) after the end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Patients may not have received the following investigational or SOC therapies within the below specified time frames prior to C1D1:

  * Denosumab or bisphosphonates within 4 weeks
  * Radiation therapy within 1 week
  * Systemic chemotherapy, including antibody drug conjugates with chemotherapy payload, within 3 weeks.
  * Immunotherapy within 3 weeks
  * Oral chemotherapy or molecularly targeted therapy within 5 half-lives of the agent.
  * Endocrine therapies do not have a required washout and may be continued until C1D1.
* Untreated brain metastases. Patients with treated brain metastases are eligible if they show no evidence of progression and are off steroids or on stable/decreasing steroid dose.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to ATI-2231.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with known HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Screening resting QTcF above 460 ms (average of triplicate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events | From baseline through 30 days after end of treatment (estimated to be 7 months)
  -Graded per CTCAE v. 5.0

SECONDARY OUTCOMES:
Changes in ATI-2231 pharmacokinetics (PK) as measured by time to peak drug concentration (Tmax) | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 day 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by elimination rate constant | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 day 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by apparent volume of distribution | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 day 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by apparent clearance | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 day 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by peak concentration (Cmax) | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 day 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by half-life (T1/2) | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by area under the curve (AUC0-24h) | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, and 24 hours post dose cycle 1 (estimated to be 1 day)
Changes in ATI-2231 pharmacokinetics (PK) as measured by area under the curve (AUC0-infinity) | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by area under the curve (AUC0-t) | Pre-dose cycle 1 day 1, 1 hour, 2 hours, 4 hours, 6 hours, 10 hours, 24 hours, 30 hours, and 48 hours post dose cycle 1 (estimated to be 2 days)
Changes in ATI-2231 pharmacokinetics (PK) as measured by peak concentration (Cmax) | Pre-dose cycle 2 day 1 (each cycle is 21 days), 1 hour, 2 hours, 4 hours, 6 hours, and 10 hours post dose cycle 2 day 1 (estimated to be 10 hours)
Changes in ATI-2231 pharmacokinetics (PK) as measured by trough concentration | Pre-dose cycle 2 day 1 (each cycle is 21 days), 1 hour, 2 hours, 4 hours, 6 hours, and 10 hours post dose cycle 2 day 1 (estimated to be 10 hours)
Changes in ATI-2231 pharmacokinetics (PK) as measured by area under the curve (AUC0-t) | Pre-dose cycle 2 day 1 (each cycle is 21 days), 1 hour, 2 hours, 4 hours, 6 hours, and 10 hours post dose cycle 2 day 1 (estimated to be 10 hours)
Changes in ATI-2231 pharmacokinetics (PK) as measured by time to peak drug concentration (Tmax) | Pre-dose cycle 2 day 1 (each cycle is 21 days), 1 hour, 2 hours, 4 hours, 6 hours, and 10 hours post dose cycle 2 day 1 (estimated to be 10 hours)
ATI-2231 pharmacokinetics (PK) as measured by trough concentration | Cycle 3 day 1 (each cycle is 21 days)
ATI-2231 pharmacokinetics (PK) as measured by trough concentration | Cycle 4 day 1 (each cycle is 21 days)
ATI-2231 pharmacokinetics (PK) as measured by trough concentration | Cycle 5 day 1 (each cycle is 21 days)
ATI-2231 pharmacokinetics (PK) as measured by trough concentration | Cycle 6 day 1 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia X Ma, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data may be shared upon request with other non-commercial researchers and the request will be reviewed by the study team after the publication.
Time Frame: After the publication
Access Criteria: Please email cynthiaxma@wustl.edu for requests.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu